CLINICAL TRIAL: NCT05684627
Title: The Application of a Fasting- Mimicking Diet in Periodontitis: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, İpek Özgü, Resident, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AkdenizU-1
Record Dates: First submitted 2022-12-20; First posted 2023-01-13 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Periodontitis
Keywords: non surgical treatment; fast-mimicking diet; systemic response; gingival crevicular fluid
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast mimicking diet group (Experimental): The patients in this group will be assigned to follow one cycle of a fasting mimicking diet (FMD) the same day after receiving the full-mouth non-surgical periodontal treatment.
  Interventions: Dietary Supplement: Fast mimicking diet group
- Normal diet group (Active Comparator): The patients in this group will be assigned to normal diet after receiving the full-mouth non-surgical periodontal treatment.
  Interventions: Procedure: Normal diet group

INTERVENTIONS:
Dietary Supplement: Fast mimicking diet group — Test group will be assigned to follow one cycle of a fasting mimicking diet the same day after receiving the full mouth non surgical periodontal treatment. The FMD program is a plant-based diet program designed to attain fasting-like effects while providing both macro- and micronutrients to minimize the burden of fasting and adverse effects. The FMD consist 5 days regimen that provides approximately 1.100 kilocalories for the first day ; approximately 750 kilocalories per day for the second to the fifth day. FMD group will need 5 visits.
  Arms: Fast mimicking diet group
Procedure: Normal diet group — Normal diet (control) group after receiving the non surgical periodontal treatment (with periodontal Gracey curettes and ultrasonic scaler) will continue with their current diet.Normal diet group will need 5 visits.
  Arms: Normal diet group

SUMMARY:
The aim of the present study is to test if a fasting mimicking diet (FMD) can influence the systemic and periodontal response following non-surgical periodontal therapy. The null hypothesis is that a FMD does not modify the local and systemic inflammatory post-treatment response.

The test group will have periodontal treatment followed by fasting mimicking diet while the control group will have the same periodontal treatment and continue with their normal diet.

Full-mouth clinical periodontal measurements including probing depth (PD), clinical attachment level (CAL), bleeding on probing (BOP), gingival index (GI) and plaque index (PI) will be recorded.Blood and GCF samples will be taken.Enzyme-linked immunosorbent assay (ELISA) will be used to determine biochemical parameters in the biological samples.

DETAILED DESCRIPTION:
This is a multi-center randomized controlled trial with internal pilot.The study protocol was approved by the Ethics Committee for the Use of Human Subjects in Research of Hatay Mustafa Kemal University. Participants will be selected from the patients who consult to the Periodontology Clinic of Akdeniz University Faculty of Dentistry. (Antalya, TURKEY).Participants will be screened by clinical staff/ investigator. We expect 20 eligible participants available per year.

The FMD program is a plant-based diet program and consists of a 5-days regimen. Test group will be assigned to follow one cycle of a fasting mimicking diet (FMD) the same day after receiving the full-mouth non-surgical periodontal treatment (NSPT). In contrast, control group after receiving the NSPT will continue with their current diet.

Patients in the test group will need 5 visits and patients in the control group will also need 5 visits.

At the screening visit, consent will be sought by the trained applicant which will be recorded through a written participant consent form detailing the complete trial procedure and an agreement checklist for each data collection method.

Visit 1 (Day -7/-10): Informed consent will be given and signed, blood and GCF samples will be collected, medical history will be checked and oral examination will be carried out including recording number of teeth and at 6 sites per tooth probing depth,recession (mm) and bleeding after probing.A very superficial prophylaxis , motivation and oral hygiene instructions will be provided.

On day 0 Morning (Visit 2) : Patients will undergo full-mouth subgingival instrumentation procedures and more detailed hygiene instruction will be reinforced. In the afternoon patients of the test group will start the FMD for 5 consecutive days.

On day 1(Visit 3) :Blood and GCF samples will be taken. Medical history, adverse events and concomitant medications will be checked.

On day 7 (Visit 4 ): Blood and GCF samples will be taken. Medical history, adverse events and concomitant medications will be checked.

On day 90±5 (visit 5): Full mouth periodontal charting measurements will be recorded. Blood and GCF sample swill be taken. Periodontal re-evaluation will be done.

The samples will be collected during the study visit from the patient by investigator, who will participate in this study. GCF Periopaper Strips will be used in the gingival crevice of the teeth. They will then be immediately measured on a calibrated Periotron 8000 electronic transducer. Once measured gcf strips for that visit will all be stored in a single 2 ml tube and pooled for further analysis.

4 ml of venous blood will be collected from the participant's arm into hemogard sterile vacutainers. The samples for serum will be centrifuged for 5 mins at 40,000 rpm then immediately divided into 1 ml aliquots and stored in a freezer at - 80°C, until required for analysis. After their initial storage, the sample will be transferred to the Microbiome and Salivary laboratories of Guy's Hospital.

Blood samples will be tested for cytokines, acute phase proteins and inflammtory markers. Gingival Crevicular Fluid will be analyzed for inflammatory mediators, antibodies, peptides and cytokines using techniques such as ELISA.

Circulating levels of IGF-1, fasting blood glucose level will be assessed to monitor the compliance of FMD.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old patients
* Periodontitis stage III-IV, grade B-C
* Systemically healthy
* Normal weight to overweight. Body mass index: 18-30
* Minimum of 24 teeth present
* Be willing and physically able to carry out all study procedures.
* Absence of hopeless teeth, acute dental conditions, teeth with endo-periodontal lesions and necrotising periodontal diseases.

Exclusion Criteria:

* Age> 70 years old
* Smokers
* Systemically compromised
* Underweight/Obese
* Pregnant
* Alcoholism
* Systemic antibiotics intake within 3 months
* Periodontal treatment in the last 12 months
* Mental illness, depression, dementia.
* Denture wearer/ presence of dental implants
* Unable or unwilling to participate in baseline or follow up examinations
* Unable or unwilling to complete the dietary intervention
* Significant food allergies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Serum CRP level | post treatment 90th day
  Crp level will be evaluated biochemically

SECONDARY OUTCOMES:
Immunological crevicular fluid analysis | baseline post treatment 1st, 7th and 90th days
  IL-6, L-1α, IL-1β, IFN-y, VEGF, FGF-β, OPG, MMP-3 and MMP-8 values will be evaluated biochemically
Clinical Attachment Level | baseline and post treatment 90 days
  The probing depth and the distance from the gingival margin to the Cement-Enamel Junction in millimeters.
Probing Pocket Depth | baseline and post treatment 90 days
  The distance from the gingival margin to the apical portion of the gingival sulcus in millimeters. Probing depths in healthy gingival sulcus normally range from 1 to 3 mm.
Bleeding on Probe | baseline and post treatment 90 days
  To accurately determine the patient's periodontal health, the dental professional will record the sulcular depths of the gingiva. Any bleeding which occurs upon probing will also be recorded. A periodontal probe is used for this test.The number of sites which bleed are used to calculate the gingival bleeding score.
Gingival Index | baseline and post treatment 90 days
  The bleeding is assessed by probing gently along the wall of soft tissue of the gingival sulcus.The GI of the individual can be obtained by adding the values of each tooth and dividing by the number of teeth examined.The probed values are scored between 0-3.
  Score 0 = Normal gingiva.
  Score 1 = Mild inflammation - slight change in color, slight edema. No bleeding on probing.
  Score 2 = Moderate inflammation - redness, edema, glazing. Bleeding on probing.
  Score 3 = Severe inflammation - marked redness and edema, ulceration. Tendency toward spontaneous bleeding.
  The GI may be used for the assessment of prevalence and severity of gingivitis in populations, groups and individuals.A score from 0.1-1.0 = mild inflammation; 1.1-2.0 = moderate inflammation from, and 2.1-3.0 signifies severe inflammation.
Plaque Index | baseline and post treatment 90 days
  The measurement of the state of oral hygiene by Silness-Löe plaque index is based on recording both soft debris and mineralized deposits on the following teeth: Missing teeth are not substituted. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3.
  0= No plaque
  1= A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  2 =Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  3 =Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Patients reported quality of life measurements | baseline and post treatment 90 days
  Patients' outcomes will be assessed by Oral Health Impact Profile-14 (OHIP-14) questionnaire which is used to evaluate the impact oral health (including functional limitations, pain, physiological discomfort, physical disability, social disability, sense of taste, diet unsatisfactory and handicap) on person's life.
  The Oral Health Impact Profile-14 (OHIP-14) was designed to assess patients' perception of the impact of oral disorders on their quality of life (QoL).
Serum CRP levels | post treatment 1st, 7th and 90th day
  Crp level will be evaluated biochemically

CONTACTS AND LOCATIONS:
Overall Officials: Kemal Ustun, Professor, Study Director — Head Of Periodontology Department; Luigi Nibali, Professor, Principal Investigator — Professor and Academic Lead for Periodontology, King's College London, Guy's Hospital; Aysegul SARI, Professor, Study Chair — Mustafa Kemal University; Giuseppe Mainas, Professor, Study Director — King's College London, Guy's Hospital
Locations (1):
- Akdeniz University Faculty of Dentistry, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mainas G, Ozgu I, Sari A, Vinciguerra M, Ide M, Ayakta BB, Ustun K, Nibali L. The application of a fasting-mimicking diet in periodontitis. A feasibility study. J Dent. 2025 May;156:105644. doi: 10.1016/j.jdent.2025.105644. Epub 2025 Feb 19. PMID 39983975